CLINICAL TRIAL: NCT03554759
Title: An Observational Cohort Study of the Use of Avatrombopag in Patients With Thrombocytopenia Associated With Chronic Liver Disease Undergoing a Procedure
Brief Title: Avatrombopag for the Treatment of Thrombocytopenia in Adults With Chronic Liver Disease Undergoing a Procedure
Status: Terminated | Type: Observational
Why Stopped: Study was terminated early due to enrollment challenges
Sponsor: Sobi, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AVA-CLD-401
Record Dates: First submitted 2018-05-22; First posted 2018-06-13 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Thrombocytopenia
Keywords: Chronic Liver Disease; Low Platelet Count
MeSH Terms: conditions — Thrombocytopenia | interventions — avatrombopag

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | US Export: No

INTERVENTIONS:
Drug: Avatrombopag — Avatrombopag dosing will be determined by the treating physician in conjunction with the FDA-approved package insert.

SUMMARY:
Phase 4 observational cohort study to characterize the treatment patterns and effects of avatrombopag use in patients with thrombocytopenia associated with chronic liver disease who are either undergoing, or have already undergone, a procedure.

DETAILED DESCRIPTION:
Data (e.g. type of procedure, platelet count, etc.) will be collected retrospectively or prospectively from patient visits occurring within approximately 7 calendar days prior to the first dose of avatrombopag, on Procedure Day, on Discharge Day, and from any clinic visit performed up to 30 days post-procedure. All treatment decisions and clinical assessments will be at the discretion of the treating physician per routine medical care and are not mandated by study design or protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patient has thrombocytopenia associated with chronic liver disease and is planned for or underwent treatment with avatrombopag prior to a procedure
* Patient provides written informed consent

Minimum Data for Retrospective Enrollment

* Platelet count from approximately 7 days prior to starting avatrombopag
* Platelet count on Procedure Day

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients ≥18 years of age who have thrombocytopenia associated with chronic liver disease and are planned for or underwent treatment with avatrombopag prior to a procedure.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Change in platelet count | Up to 8 days after the last dose of avatrombopag.

SECONDARY OUTCOMES:
Proportion of patients who received a platelet transfusion | From the first dose of avatrombopag to up to 15 days after the last dose of avatrombopag
Occurrence of adverse events | From the first dose of avatrombopag to up to 30 days after the last dose of avatrombopag

CONTACTS AND LOCATIONS:
Locations (40):
- United States (40):
  - Dova Site, Chandler, Arizona
  - Dova Site, Lancaster, California
  - Dova Study Site, Los Angeles, California
  - Dova Site, Palm Springs, California
  - Dova Study Site, Pasadena, California
  - Dova Study Site, San Clemente, California
  - Dova Study Site, San Diego, California
  - Dova Study Site, Aurora, Colorado
  - Dova Study Site, Englewood, Colorado
  - Dova Study Site, Gainesville, Florida
  - Dova Study Site, Miami, Florida
  - Dova Study Site, Atlanta, Georgia
  - Dova Study Site, Topeka, Kansas
  - Dova Study Site, Louisville, Kentucky
  - Dova Study Site, Baltimore, Maryland
  - Dova Study Site, Boston, Massachusetts
  - Dova Study Site, Burlington, Massachusetts
  - Dova Study Site, Worcester, Massachusetts
  - Dova Study Site, Ann Arbor, Michigan
  - Dova Study Site, Detroit, Michigan
  - Dova Site, Jackson, Mississippi
  - Dova Study Site, New Brunswick, New Jersey
  - Dova Study Site, Manhasset, New York
  - Dova Study Site, New York, New York
  - Dova Study Site, The Bronx, New York
  - Dova Study Site, Durham, North Carolina
  - Dova Study Site, Cleveland, Ohio
  - Dova Study Site, Columbus, Ohio
  - Dova Study Site, Flourtown, Pennsylvania
  - Dova Site, Philadelphia, Pennsylvania
  - Dova Study Site, Pittsburgh, Pennsylvania
  - Dova Study Site, Johnson City, Tennessee
  - Dova Study Site, Memphis, Tennessee
  - Dova Study Site, Union City, Tennessee
  - Dova Study Site, Dallas, Texas
  - Dova Study Site, Houston, Texas
  - Dova Study Site, Charlottesville, Virginia
  - Dova Study Site, Richmond, Virginia
  - Dova Study SIte, Roanoke, Virginia
  - Dova Study Site, Milwaukee, Wisconsin